CLINICAL TRIAL: NCT02315833
Title: The Efficacy of L-cysteine in Prevention of Headache Attacks in Migraine Patients. Randomized Intervention Trial With a Medical Device (Acetium®Capsules)
Brief Title: The Efficacy of L-cysteine in Prevention of Headache Attacks in Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biohit Oyj (Industry)
Collaborators: The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-MIGPREV-1
Record Dates: First submitted 2014-12-04; First posted 2014-12-12 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Migraine
Keywords: Migraine; Aura
MeSH Terms: conditions — Migraine Disorders; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetium (Experimental): Patient will administer Acetium capsules (100mg l-cysteine) twice a day for three months
  Interventions: Drug: Acetium
- Placebo (Placebo Comparator): Patient will administer placebo capsules twice a day for three months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetium — Capsule for oral administration contains L-cysteine 100mg
  Other Names: Acetium capsule
  Arms: Acetium
Drug: Placebo — A placebo capsule matching Acetium for oral administration.
  Other Names: Acetium capsule placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to validate the novel hypothesis that daily use of L-cysteine (Acetium® capsules) is an effective means to decrease the frequency of (or completely abort) the headache attacks in migraine patients.

DETAILED DESCRIPTION:
Background: Globally, 15% of the population is affected by migraines at some point in their life-time. Pprophylactic treatment of migraines is an important part of the total management of migraine patients, having twofold goals: i) to reduce the frequency, painfulness, and/or duration of migraines, and ii) to increase the effectiveness of abortive therapy. During the past several decades, a large number of optional modalities have been tested as preventive measures of migraine attacks. Not unexpectedly, the effects of any such preventive therapies are highly variable, and in many patients, the attack frequency is not under satisfactory control. Many of these drugs also have untoward side effects that offset their potential benefits.

Recently, spontaneous case testimonials were received by Biohit Oyj from migraine patients, reporting that our new medical device, Acetium™ capsule (containing 100mg L-cysteine, developed for inactivation of acetaldehyde in the stomach contents after alcohol intake), proved to be highly effective against migraine attacks. Their headache attacks disappeared almost immediately after onset of L-cysteine administration, all of them remaining in complete remission for several months up to several years by now.

These spontaneous testimonials prompted us to formulate a novel study hypothesis that could possibly explain these dramatic effects of L-cysteine in migraine prevention, to be tested in this RCT. This novel hypothesis is starting from the fact that, swelling and dilatation of cerebral blood vessels is necessary to provoke the attack in this vascular-type of headache.

It is known that Nitric Oxide (NO) is the final trigger of migraine attack, operating through phosphorylated protein kinase G (PKG) and Ca2+ channels, slowing the influx of calcium into the cell, which leads to smooth muscle relaxation and vasodilation. Histamine is a potent inducer of NO Synthase, making NO available locally on the vasculature, acting through endothelial H1-receptors. Histamine is synthesized from histidine in tissue mast cells, which are ubiquitous cells and their activation e.g. in the meninges has long been suspected to be involved in generating migraine headaches. Finally, one of the potent liberators of histamine from the mast cells is acetaldehyde, which, in turn, is effectively inactivated by L-cysteine (Acetium capsule). This led us to rational that by eliminating acetaldehyde in the stomach, L-cysteine could block (or reduce below the threshold levels) histamine liberation from the tissue mast cells and ECL cells in the stomach, thus arresting its multitude of functions, of which vasodilatation is critically involved in the migraine attack.

Objective: To validate the novel hypothesis that daily use of L-cysteine is an effective means to decrease the frequency of (or completely abort) the headache attacks in migraine patients.

Study design: A double-blind, randomized placebo-controlled multi-centre trial comparing Acetium capsules (100mg L-cysteine, twice a day) and placebo in prevention of migraine attacks during a 3-month trial period. A cohort of 200 voluntary subjects (women and men, with aural or non-aural migraine) are invited through the Finnish Migraine Association (FMA), to participate in the study. To be eligible, the subjects should: i) have the attack frequency of 2-8 times per month, ii) have had migraine for at least 1 year, iii) have the onset of their migraine before 50 years of age, iv) be between 18 and 65 years of age, and v) have a minimum of co-morbidity. Eligible patients are allowed (if they want) to continue their current migraine prophylactic medication prior to study entry. Before enrolment in the cohort, all subjects are requested to sign a written consent. The study protocol will be subjected for approval by the Regional Committee on Medical Research Ethics (HUS).

Methods: A 3-month retrospective history and 1-month prospective baseline (run-in) period is used to assess the baseline attack frequency. The study setting is actually triple-blinded (participant-blind, investigator-blind, sponsor-blind). Placebo preparation with design and package identical to the test preparation will be used. Parallel group design instead of cross-over design is used. Randomization will be performed using a random number generator, with blocks size of 4, and creating unique randomization codes for each subject. The stratified randomization is based on the attack frequency is used as the stratification variable, using 4 attacks per month as the cut-off for low-and high frequency.

The treatment period in both study arms will be 3 months. The participants should use (and accurately report) their usual symptomatic or acute treatment, because not anticipated to interfere with the study medication. During the 3-month treatment period, participants will be evaluated at monthly intervals by the study coordinator. As determined by the final study compliance, data analyses might be necessary separately for i) Per Protocol (PePr), and ii) Intention-to-treat (ITT) groups.

In addition to the baseline assessment of attack frequency, each subject will be requested to fill in a structured Questionnaire recoding their detailed migraine history and other pertinent data on potential triggers, to be used as covariates in multivariate analysis. The headache diary is the main research tool used to monitor the efficacy of the test preparations, recording all predefined assessment measures (efficacy, tolerability and safety). These diaries are submitted to the study monitor on each FU visit, to confirm the compliance.

In statistical analysis, both conventional techniques (e.g. non-parametric paired-samples and non-paired samples t-test), and more sophisticated methods will be used. The latter include i) life-table methods like Kaplan-Meier and Cox proportional hazards regression, as well as ii) generalized linear models (GEE and panel Poisson) and as a new technique in migraine RCTs, a competing risks regression, to model the natural outcomes of migraine during the intervention. This study (n=100 per study arm) is adequately powered (Type II error 0.80, type I error 0.05) to detect a true difference in attack frequency between 4 attacks/month in the placebo and 2.4 attacks/month in the Acetium arm, i.e., the difference in effect size of 1.6 attacks. Given that the study subjects are selected among patients with 2-8 monthly attacks, there figures seem reasonable estimates for the basis of these power calculations.

Specific aims: The null hypothesis of the study implicates that l-cysteine is no better than placebo in migraine prophylaxis during the intervention period of 3 months. Rejection or not of the null hypothesis is based on comparison of the two arms for two primary study endpoints and (to lesser extent) for a series of secondary endpoints. The two primary study endpoints (efficacy measures) are: a) Number of migraine attacks (NMA) per evaluation interval (1 month), and ii) Number of migraine days (NMD) per evaluation period. Potentially useful secondary endpoints include: i) Intensity of headache (4-tier nominal scale); ii) Attack duration in hours (potentially biased by treatment); iii) Drug consumption for symptomatic or acute treatment (NMDs treated with abortive agents and the number of drug administrations for acute therapy); iv) Patients' preferences and satisfaction; v) Responder rate (proportion of study subjects with >50% improvement in NMA or NMD, as compared to baseline values).

Study execution and time table: Meanwhile the final protocol is under evaluation for ethical approval by HUS, preparatory measures have been taken by informing the FMA about the planned study and asking their co-operation in encouraging the interested migraine patients to contact the study coordinator. Given the preliminary interest shown by the FMA, we are optimistic that the required cohort of volunteers can be enrolled within a short time, most likely by the end of 2013. Because each study subject shall complete only a 3-month trial period, preceded by 1-month run-in time, we expect that the study will be completed during the second half of 2014.

Impact of the study: Given that L-cysteine is a natural (semi-essential) amino acid, converted to inert substance (MTCA) in the alimentary tract, it would comprise an ideal means to conduct migraine prophylaxis for years, without concern about the side effects that are inherent to many of the current treatment modalities. If the efficacy is proved in this formal RCT, the concept of using Acetium capsules in prophylactic treatment of migraines would represent a major step forward in a better clinical control of these frequently intractable syndromes.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years male/female
* subjects should report migraine attacks with the frequency of 2-8 times per month, and with less than 15 migraine days (NMD) per month. To be calculated as a separate attack, there should be at least 48h of freedom from headache between the two attacks of migraine.
* migraine with or without aura has been present for at least 1 year prior to entering into the study
* subjects to be enrolled should report the onset of their migraine before 50 years of age

Exclusion Criteria:

* patients who meet the International Classification of Headache Disorders II criteria for medication overuse
* patients who have taken anti-psychotics or anti-depressant medications during the previous 3 months
* patients who abuse alcohol or other drugs
* patients resistant to all acute migraine drugs optimally prescribed
* potentially fertile and sexually active women who do not practise contraception
* other acute or chronic pain disorders
* severe psychiatric disease
* infection
* malignancy
* short life expectancy
* cardiovascular disease
* cerebrovascular disease
* uncontrolled hypertension
* degenerative central nervous system diseases
* pregnant and lactating women
* regular users of Acetium capsules for other indications
* persons suffering from renal dysfunction or cystinuria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-12-17 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Number of migraine attacks (NMA) per evaluation interval | 3 months
  The frequency of headache attacks during the entire treatment period (3 months) is compared with the baseline frequencies, to disclose the differences in efficacy measures between the two arms.

SECONDARY OUTCOMES:
Number of migraine days (NMD) per evaluation period | 3 months
  The frequency of headache days during the entire treatment period (3 months) is compared with the baseline frequencies, to disclose the differences in efficacy measures between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Syrjänen, MD, PhD, Study Chair — Biohit Oyj; Mikko Kallela, MD, PhD, Principal Investigator — Helsingin Päänsärkykeskus Oy
Locations (7):
- Estonia (2):
  - Confido Privat Medical Clinic, Tallinn
  - Tartu University Hospital, Neurology Clinic, Tartu
- Finland (5):
  - Terveystalo, Kamppi, Helsinki
  - Lääkärikeskus Aava, Helsingin Päänsärkykeskus Oy, Helsinki
  - Terveystalo, Jyväskylä, Jyväskylä
  - Terveystalo, Oulu, Oulu
  - Terveystalo, Turku, Turku

IPD SHARING:
Plan to Share IPD: No